CLINICAL TRIAL: NCT07134933
Title: The Effects of Erector Spinae Plane Block on Pain Scores and Patient Experience in Unilateral Breast Cancer Surgery: A Prospective, Randomized Clinical Trial
Brief Title: The Effects of Erector Spinae Plane Block on Pain Scores in Unilateral Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Mukadder Sanli, Associate professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ESP Block
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Erector Spinae Plane Block
Keywords: Erector spinae plane block; patient satisfaction; breast surgery; postoperative analgesia
MeSH Terms: conditions — Patient Satisfaction | interventions — Parapsychology

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): The group with ESP block was defined as Group 1. The ESP block was performed unilaterally in the direction of the surgery.
  Interventions: Procedure: ESP (erector spinae plane)block
- Group II (No Intervention): The group without ESP block was defined as Group II.

INTERVENTIONS:
Procedure: ESP (erector spinae plane)block — The ESP block was performed unilaterally in the direction of the surgery by the same anesthetist. Blocks were performed using an Esaote ultrasound device (Esaote My Lab 6 US machine, Florence, Italy), a multifrequency convex probe (1-8 MHz), and a 22-gauge, 50 mm facet needle (B. Braun Sonoplex, Melsungen, Germany). The block needle was placed at the level of the T4 spinal process using the in-plane approach, approximately 3 cm lateral to the T4 spinous process in the parasagittal plane. After visualizing the transverse process with the in-plane approach, the 50 mm facet needle (B. Braun Sonoplex, Melsungen, Germany) was inserted through the skin, and a test dose of 1 ml of 0.9% NaCl was injected between the fascia of the trapezius, rhomboid, and erector spinae muscles and the transverse vertebral process to confirm the location. A total of 20 ml of 0.5% bupivacaine was used as a local anesthetic.
  Arms: Group I

SUMMARY:
The high incidence of breast cancer is increasing the need for oncologic breast surgery. The optimal acute postoperative pain management after breast surgery is not yet clear. The erector spinae plane block (ESPB) is a newer and may be potentially safer alternative other regional analgesia techniques. We will investigate the effectiveness of ESP for managing acute pain after breast cancer surgery. Patients will randomise to receive either ESP block (Group1)or no ESP block (Group II). The primary outcome is postoperative pain scores used Visual Analog Scale (VAS), and the secondary outcomes include intraoperative opioid consumption postoperative total opioid consumption and patient satisfaction.

DETAILED DESCRIPTION:
Anesthesia induction was achieved with propofol (2-3 mg kg-1), fentanyl (2 mcg kg-1), and rocuronium (0.6 mg kg-1). Anesthesia was maintained with Total intravenous anesthesia (TIVA) used remifentanil (0.25-0.5 mcg kg-1 min-1) and propofol (150 mcg kg-1 min-1). During maintenance, a fresh gas flow of 3 L with a mixture of 50% oxygen and 50% air was used. The BIS value was kept between 30-50.

Patients were divided into two groups according to a computer-based simple randomization method. Those who received a preoperative ESP block at the T4 vertebra level under ultrasound guidance were designated as Group I, while those who underwent surgery without the block were designated as Group II.

The ESP block was performed unilaterally in the direction of the surgery by the same anesthetist. Blocks were performed using an Esaote ultrasound device (Esaote My Lab 6 US machine, Florence, Italy), a multifrequency convex probe (1-8 MHz), and a 22-gauge, 50 mm facet needle (B. Braun Sonoplex, Melsungen, Germany) The block needle was placed at the level of the T4 spinal process using the in-plane approach, approximately 3 cm lateral to the T4 spinous process in the parasagittal plane. After visualizing the transverse process with the in-plane approach, the 50 mm facet needle (B. Braun Sonoplex, Melsungen, Germany) was inserted through the skin, and a test dose of 1 ml of 0.9% NaCl was injected between the fascia of the trapezius, rhomboid, and erector spinae muscles and the transverse vertebral process to confirm the location. A total of 20 ml of 0.5% bupivacaine was used as a local anesthetic. The cranial and caudal spread of the local anesthetic was monitored.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* the patients who undergone unilateral surgery due to breast tumors

Exclusion Criteria:

* obesity (body mass index> 35 kg/m²)
* infection at the needle entry site,
* known allergy history to the medications to be used,
* coagulopathy
* a history of opioid use

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since patients were required to undergo breast surgery, only female gender was included in the study.
Enrollment: 68 (Actual)
Dates: Start 2018-12-25 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-04-20 (Actual)

PRIMARY OUTCOMES:
Remifentanil Consumption | From beginning of anesthesia to finished the surgery
  The primary aim of our study was to compare perioperative remifentanil consumption between Group I patients who received a preoperative ESP block and Group II patients who underwent surgery without the block.

SECONDARY OUTCOMES:
postoperative morphine consumption | from the end of the surgery to 24 hours of postoperative
  After extubation, a patient-controlled analgesia device containing morphine (0.5 mg/ml, 1 mg bolus, 8-minute lockout interval, maximum dose of 6 mg in 1 hour) was installed. The amount of morphine consumed in the postoperative 24 hours was measured.
The VAS scores | from the end of the surgery to 24 hours of postoperative
  Postoperative pain assessment was conducted using the Visual Analog Scale (VAS), where 0 indicates no pain and 10 indicates unbearable pain) at rest and during movement at the 5, 15, 30, and 60 minutes, as well as at 2, 4, 6, 8, 16, and 24 hours post-surgery.
patient satisfaction | at the 24th postoperative hour
  a four-point patient satisfaction score (1: poor, 2: fair, 3: good, 4: excellent) were evaluated by an anesthetist who was unaware of the study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mukadder Sanli, Associate Professor, Study Chair — Inonu University
Locations (1):
- İnonu University Medicine Faculty Turgut ozal Medical Center, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We do not want our data to be used by others.

REFERENCES:
- [Background] Wick EC, Grant MC, Wu CL. Postoperative Multimodal Analgesia Pain Management With Nonopioid Analgesics and Techniques: A Review. JAMA Surg. 2017 Jul 1;152(7):691-697. doi: 10.1001/jamasurg.2017.0898. PMID 28564673